CLINICAL TRIAL: NCT04936620
Title: Duroplasty for Injured Cervical Spinal Cord With Uncontrolled Swelling
Acronym: DISCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other); St. Mary's University, Twickenham (Other); University of Bristol (Other); Ohio State University (Other); University of Cambridge (Other); University of Oxford (Other); Buckinghamshire Healthcare NHS Trust (Other); Paracelsus Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021.0056; 25573423 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries
Keywords: Decompression, surgical; Neurosurgery; Paralysis
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Intervention Model Description: Phase III clinical trial: randomised, controlled, double blind, multi-centre, superiority
  + Optional mechanistic study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants, some care providers (ie: physiotherapists) and outcome assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duroplasty (Active Comparator): Duroplasty (includes Surgery with Laminectomy)
  Interventions: Procedure: Duroplasty; Procedure: Spinal surgery
- No duroplasty (Active Comparator): No duroplasty (but includes surgery with Laminectomy)
  Interventions: Procedure: Spinal surgery

INTERVENTIONS:
Procedure: Duroplasty — Expansion Duroplasty
  Arms: Duroplasty
Procedure: Spinal surgery — Spinal surgery including laminectomy

SUMMARY:
QUESTION. Does duroplasty improve outcome after spinal cord injury?

WHAT DO WE STUDY? We will investigate whether performing a surgical procedure called duroplasty improves outcomes after spinal cord injury.

WHY SPINAL CORD INJURY? Spinal cord injury is a devastating condition that causes permanent disability such as paralysis, numbness and loss of bladder and bowel control. Currently, there are no treatments shown to improve outcome after spinal cord injury.

WHAT IS DUROPLASTY? Duroplasty is an operation that involves opening the tough membrane around the cord, called the dura, and stitching a patch of artificial dura to expand the space around the swollen cord.

WHY IS DUROPLASTY BEING STUDIED? Based on our preliminary evidence, we think that the dura causes cord pressure after injury. We have shown in a small study of patients that performing this operation safely and effectively reduces pressure on the injured cord.

WHO IS ELIGIBLE? Adult patients with severe spinal cord injuries in the neck who will have surgery within 72 hours.

WHAT TREATMENT? Those who agree to take part will be allocated by chance (like tossing a coin) to standard treatment or standard treatment plus duroplasty. Some patients will also be asked to take part in a smaller study that involves placing probes at the injury site.

WHERE? We will recruit patients from U.K. Major Trauma Centres. Most assessments will be done in U.K. Spinal Injury Centres. Later on, we may recruit from overseas.

HOW LONG? We aim to recruit 222 - 260 patients over 4 years. Patients will be followed up for a year.

WHAT DO WE ASSESS? Patients will be assessed (using questionnaires and by examination) how well they can use their hands, walk, control their bladder and bowel and their quality of life. Some of these assessments will be repeated at 3, 6 and 12 months after surgery.

WHAT IS THE OPTIONAL MECHANISTIC STUDY? DISCUS includes an optional study for at least 50 patients who will take part in the randomised controlled trial. The aim of the mechanistic study is to determine how duroplasty improves outcome, i.e. whether duroplasty reduces cord compression, improves blood flow to the injured cord perfusion, improves cord metabolism and reduces cord inflammation.

WHAT IS THE OPTIONAL INFORMATION STUDY? For the first two years, a study called QuinteT Recruitment Intervention (QRI) is designed to optimise patient recruitment and informed consent in the trauma setting.

DETAILED DESCRIPTION:
RESEARCH QUESTION: After severe traumatic spinal cord injury (TSCI), does the addition of dural decompression to bony decompression (includes laminectomy) improve muscle strength in the limbs at 6 months, compared with bony decompression alone? BACKGROUND: TSCI is a devastating condition that affects about 1,000 people in the UK annually. Most remain disabled, tetraplegic or wheelchair bound and are dependent on carers with significant cost to patients, carers and the NHS. Surgery aims to reduce spinal deformity, stabilise the spine and achieve bony decompression of the cord. To date, no treatments have been shown to improve outcome.

AIMS / OBJECTIVES: The primary aim is to determine if, in patients with acute, severe TSCI, the addition of dural decompression to bony decompression improves muscle strength. We hypothesise that, after TSCI, the cord swells and is compressed against the dura. Secondary objectives are to assess patient impact i.e. functional outcomes, health related quality of life (HRQoL), complication rates and mortality. Mechanistic sub-studies aim to determine if the addition of duroplasty improves cord perfusion, reduces cord ischaemia and cord inflammation.

METHODS: This is a prospective, phase III, multicentre randomised controlled trial (RCT). We aim to recruit 222 adults with acute, severe cervical TSCI (American spinal injuries association Impairment Scale (AIS) grade A, B or C) who will be randomised 1:1 to undergo bony decompression alone versus bony decompression with duroplasty. Patients and assessors will be blinded to study arm. The primary outcome is change in AIS motor score (AMS) at 6 months compared with admission (Delta-AMS); secondary outcomes will assess function (grasp, walking, urinary + anal sphincters), HRQoL, complications, need for further surgery and mortality, assessed at baseline, 3 months, 6 months and 12 months from randomisation. A subgroup of 50 patients (25 per arm) will also have observational monitoring from the injury site using a pressure probe (intraspinal pressure ISP, spinal cord perfusion pressure SCPP) and microdialysis (MD) catheter (cord metabolism: tissue glucose, lactate, pyruvate, lactate-to-pyruvate ratio (LPR), glutamate, glycerol); cord inflammation: tissue chemokines/cytokines. Patients will be recruited from the 26 UK major trauma centres (MTCs).

TIMELINES FOR DELIVERY: The initial study duration was 72 months and includes 6 months set-up, 48 months recruitment, 12 months to complete follow-up and 6 months for data analysis and final reporting of results. There will be a formal stop/go review at month 15 (after 9 months of recruitment) to ensure a minimum of 4 sites have been opened and 8 patients randomised. If these targets are met, the trial will recruit for a further 36 months. Data from the pilot will be included in the final analysis. Recruitment has been extended to end on 30 June 2027.

ANTICIPATED IMPACT AND DISSEMINATION: It is anticipated that the addition of duroplasty to standard of care will improve muscle strength in patients; this has obvious benefits for patients and their carers as well as substantial gains for the NHS and society including economic implications. If this RCT shows that the addition of duroplasty to standard treatment is beneficial, it is anticipated that duroplasty will become standard NHS care in all 26 UK MTCs. Participants will be informed of study findings via the Surgical Intervention Trials Unit (SITU) website and the Spinal Injuries Association (SIA).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16 years
2. Severe cervical (C2 - T1) traumatic spinal cord injury (AIS grade A-C)
3. Deemed to require and be suitable for surgery that includes laminectomy by local surgeon
4. Surgery within 72 hours of traumatic spinal cord injury
5. Able to provide informed consent or consultee declaration or proxy consent.

Exclusion Criteria:

1. Dural tear due to traumatic spinal cord injury
2. Life-limiting or rehabilitation-restricting co-morbidities
3. Thoracic or lumbar traumatic spinal cord injury
4. Other central nervous system disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in AIS motor score | 6 months versus baseline
  Change in American Spinal Injury Association Impairment Scale total limb motor score at 6 months

SECONDARY OUTCOMES:
Change in AIS light touch score | 6 months versus baseline
  Change in American Spinal Injury Association Impairment Scale total light touch sensory score
Change in AIS pin prick score | 6 months versus baseline
  Change in American Spinal Injury Association Impairment Scale total pin prick sensory score
Change in AIS grade | 6 months versus baseline
  Change in American Spinal Injury Association grade
CUE-Q | 6 months
  Capabilities of upper extremity-questionnaire (CUE-Q)
Grip strength | 6 months
  Hand grip strength assessed with dynamometer
WISCI II | 6 months
  Walking Index for Spinal Cord Injury version ii
SCIM III | 6 months
  Spinal Cord Independence Measure version III
SF-36 | 6 months, 12 months
  Short Form survey 36
Spinal re-operations | 12 months
  Number of reoperations on spine
Adverse events | 12 months
  Procedure Specific complications and adverse events
Mortality | 12 months
  Mortality
Length of hospital stay | 12 months
  Length of hospital stay
MRI | 2 weeks, 6 months
  Magnetic resonance imaging of cervical spine
Injury site physiology and metabolism (optional) | Up to 5 days after surgery
  Optional mechanistic study: Mean daily intraspinal pressure, spinal cord perfusion pressure, tissue glucose, lactate, pyruvate, glycerol, glutamate, cytokines measured from the injury site

CONTACTS AND LOCATIONS:
Overall Officials: Marios C Papadopoulos, Principal Investigator — St George's, University of London, U.K.; Samira Saadoun, Principal Investigator — St George's, University of London, U.K.
Locations (33):
- Austria (4):
  - Universität Klinik für Neurochirurgie, Innsbruck
  - Kepler University Hospital, Linz
  - University Hospital Salzburg, Salzburg
  - St Polten University Hospital, Sankt Pölten
- UZ Leuven, Leuven, Belgium
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China
- Masaryk Hospital, Ústí nad Labem, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- Kuopio University Hospital, Kuopio, Finland
- BG Unfallklinik Frankfurt am Main, Frankfurt, Germany
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Centre, Jerusalem
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- 12 de Octubre University Hospital, Madrid, Spain
- Skåne University Hospital, Lund, Sweden
- United Kingdom (18):
  - National Spinal Injuries Centre, Aylesbury
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - The Walton Centre, Liverpool
  - St George's Hospital, London
  - St Mary's Hospital, London
  - The London Spinal Cord Injury Centre, London
  - The Royal London Hospital, London
  - Queen's Medical Centre, Nottingham
  - Midlands Centre for Spinal Injuries,, Oswestry
  - Salford Royal, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - North West Regional Spinal Injuries Centre, Southport
  - Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Appropriately anonymised datasets from our sponsored research will be made available for further analysis wherever possible under our Research Data Management policy:
  https://www.sgul.ac.uk/about/governance/policies/research-data-management
Supporting Information: Study Protocol, CSR
Time Frame: Publications on this study will be available form PubMed, Study website and other publicly accessible resources.
Access Criteria: Specific requests for data sharing should be directed to sponsor St George's University London.
URL: https://www.sgul.ac.uk/about/governance/policies/research-data-management

REFERENCES:
- [Background] Saadoun S, Asif H, Papadopoulos MC. The concepts of Intra Spinal Pressure (ISP), Intra Thecal Pressure (ITP), and Spinal Cord Perfusion Pressure (SCPP) in acute, severe traumatic spinal cord injury: Narrative review. Brain Spine. 2024 Oct 16;4:103919. doi: 10.1016/j.bas.2024.103919. eCollection 2024. PMID 39654909
- [Background] Saadoun S, Grassner L, Belci M, Cook J, Knight R, Davies L, Asif H, Visagan R, Gallagher MJ, Thome C, Hutchinson PJ, Zoumprouli A, Wade J, Farrar N, Papadopoulos MC. Duroplasty for injured cervical spinal cord with uncontrolled swelling: protocol of the DISCUS randomized controlled trial. Trials. 2023 Aug 7;24(1):497. doi: 10.1186/s13063-023-07454-2. PMID 37550727
- [Background] Werndle MC, Saadoun S, Phang I, Czosnyka M, Varsos GV, Czosnyka ZH, Smielewski P, Jamous A, Bell BA, Zoumprouli A, Papadopoulos MC. Monitoring of spinal cord perfusion pressure in acute spinal cord injury: initial findings of the injured spinal cord pressure evaluation study*. Crit Care Med. 2014 Mar;42(3):646-55. doi: 10.1097/CCM.0000000000000028. PMID 24231762
- [Background] Phang I, Werndle MC, Saadoun S, Varsos G, Czosnyka M, Zoumprouli A, Papadopoulos MC. Expansion duroplasty improves intraspinal pressure, spinal cord perfusion pressure, and vascular pressure reactivity index in patients with traumatic spinal cord injury: injured spinal cord pressure evaluation study. J Neurotrauma. 2015 Jun 15;32(12):865-74. doi: 10.1089/neu.2014.3668. Epub 2015 May 4. PMID 25705999
- [Background] Phang I, Zoumprouli A, Papadopoulos MC, Saadoun S. Microdialysis to Optimize Cord Perfusion and Drug Delivery in Spinal Cord Injury. Ann Neurol. 2016 Oct;80(4):522-31. doi: 10.1002/ana.24750. Epub 2016 Aug 19. PMID 27463064
- [Background] Saadoun S, Papadopoulos MC. Acute, Severe Traumatic Spinal Cord Injury: Monitoring from the Injury Site and Expansion Duraplasty. Neurosurg Clin N Am. 2021 Jul;32(3):365-376. doi: 10.1016/j.nec.2021.03.008. Epub 2021 May 7. PMID 34053724
- See also: DISCUS NIHR Research Award — https://fundingawards.nihr.ac.uk/award/NIHR130048
- See also: DISCUS ISRCTN registry — https://doi.org/10.1186/ISRCTN25573423
- See also: DISCUS website — https://discus.octru.ox.ac.uk/discus/welcome-to-the-discus-trial
- See also: Wings for Life — https://www.wingsforlife.com/uk/research/discus-study-duroplasty-for-the-injured-cervical-spinal-cord-with-uncontrolled-swelling1

DOCUMENTS (2):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04936620/Prot_002.pdf
  • Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT04936620/ICF_003.pdf